CLINICAL TRIAL: NCT04138147
Title: Efficacy of Superficial Cervical Plexus Block Versus Cervical Retrolaminar Block Both Combined With Auriculotemporal Nerve Block in Parotid Surgeries
Brief Title: Superficial Cervical Plexus Versus Retrolaminar Block in Parotid Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MD/19.03.162
Record Dates: First submitted 2019-10-21; First posted 2019-10-24 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Supportive Care
Keywords: Cervical plexus,; Retrolaminar,; Auriculotemporal,; Parotid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Superficial cervical plexus with auriculotemporal nerve blocks (Active Comparator)
  Interventions: Procedure: Superficial cervical plexus with auriculotemporal nerve blocks
- Cervical retrolaminar with auriculotemporal nerve blocks (Experimental)
  Interventions: Procedure: Cervical retrolaminar with auriculotemporal nerve blocks

INTERVENTIONS:
Procedure: Superficial cervical plexus with auriculotemporal nerve blocks — Superficial cervical plexus block using 10 ml bupivacaine 0.5%. Auriculotemporal nerve block using 3 ml bupivacaine 0.5%.
  Arms: Superficial cervical plexus with auriculotemporal nerve blocks
Procedure: Cervical retrolaminar with auriculotemporal nerve blocks — Cervical retrolaminar block using 10 ml bupivacaine 0.5%. Auriculotemporal nerve block using 3 ml bupivacaine 0.5%.
  Arms: Cervical retrolaminar with auriculotemporal nerve blocks

SUMMARY:
The parotid gland receives sensory and autonomic innervation. Sensory innervation is supplied by the auriculotemporal nerve (gland) and the great auricular nerve (fascia). The parasympathetic innervation to the parotid gland begins with the glossopharyngeal nerve. This nerve synapses with the otic ganglion. The auriculotemporal nerve then carries parasympathetic fibers from the otic ganglion to the parotid gland. Parasympathetic stimulation increase saliva production. Sympathetic innervation from the superior cervical ganglion, part of the paravertebral chain

DETAILED DESCRIPTION:
Detailed Description:

The aim of this study will be comparing efficacy of superficial cervical plexus block with cervical retro laminar block both combined with auriculotemporal nerve block in parotid surgeries.

Technique of ultrasound guided auriculotemporal nerve block:

The patient will be placed in a supine position with each side facing up. The temporomandibular joint will be identified after palpitation. A high frequency linear ultrasound transducer (7-12 megahertz) will be attached to ultrasound machine (SIEMENS ACUSON P300, Germany) will be placed between the tragus and temporomandibular joint. Color Doppler imaging will be used to identify the superficial temporal artery. The injection needle will be inserted anterior to the tragus posterior to the temporal artery (out-of-plane approach) 1 to 1.5 cm till reaching the periosteum. The reason of out-of-plane approach is that the superficial temporal artery is in the needle entry of in-plane procedure during auriculo-temporal nerve block. Following negative aspiration local anesthetic will be injected in fractionated doses following intermittent aspiration.

Technique of ultrasound guided superficial cervical plexus block:

Standard precautions for the ultrasound guided nerve blocks performance will be done which include standard monitoring, the skin overlying the injection site will be free of signs of infection and after proper skin sterilization with an antiseptic solution and the probe surface in contact with the skin will be covered with a sterile adhesive dressing Patients will be in the supine position with the head turned slightly away from the side to be blocked to facilitate operator access. The anesthesiologist will be at the patient's side at the level of the shoulder. Posterior in-plane approach to the superficial cervical plexus block will be done. In this approach, a high-frequency linear transducer (7-12 Megahertz) will be attached to ultrasound machine (SIEMENS ACUSON P300), the transducer will be placed in a transverse orientation across the neck with the probe marker facing medial (toward the thyroid cartilage). A 22-gauge needle will then be inserted at the posterior border of the sternocleidomastoid muscle at the level of the cricoid cartilage and advanced underneath the muscle belly toward the carotid artery. The needle tip will be positioned to inject local anesthetic deep to the sternocleidomastoid muscle along its tapering posterolateral border but superficial to the prevertebral fascia. Deeper injection should be avoided because it can result in a deep cervical plexus block. As much as 10 ml of local anesthetic will be used for this block.

Technique of ultrasound guided cervical retrolaminar block:

The patients will be in the lateral position. Patient neck will be slightly flexed forward, the anesthesiologist will stand behind the patient. Firstly, landmark will be the identification of cervical vertebrae number 7 as it is the largest and most prominent spinous process by palpation in axial plane. Then the high-frequency linear transducer (7-12 Megahertz) which attach to ultrasound machine (SIEMENS ACUSON P300), Ultrasound scanning will be performed while the probe in transverse position in the mid sagittal plane of cervical vertebrae number 7 spinous process. Then counting up the spinous processes till reaching the spinous process of cervical vertebrae number 4 and then the probe will be moved laterally 1 cm to image the left or right muscles. Identification of the echogenic (bright, reflective) laminae will be seen, above it muscles will be imaged. The splenius capitis lies deep to the trapezius and is a broad, flat muscle. The semispinalis capitis will be easily recognized as a long, strap-like muscle divided into 2 sections by an aponeurotic intersection. The deep neck muscle group has a distinctive tear drop shape (semispinalis cervicis, multifidus, and rotatores).

An in-plane approach by using a 22 gauge, 50 mm, echogenic needle. The needle will be introduced to reach the lamina. After negative aspiration the local anesthetic will be injected through the needle under real-time ultrasound visualization. The criteria for assessment of correct spread of the injectate will creating a plane/hypo-echoic.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status grade I and grade II.
* Elective parotid surgery.

Exclusion Criteria:

* Patient refusal.
* Coagulopathy.
* Psychiatric diseases.
* Local skin infection and sepsis at site of the block.
* Known intolerance to the study drugs.
* Body Mass Index > 40 Kg/m2.
* Central or peripheral neurological disease.
* Previous neck surgery.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2019-11-20 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The time of first analgesic request post-operative. | 24 hours postoperative.
  The time of first analgesic request in hours.

SECONDARY OUTCOMES:
Total post-operative opioid requirement. | 24 hours postoperative.
  Total post-operative morphine requirement in milligrams..
The number of patients required rescue post-operative opioid analgesia.. | 24 hours postoperative.
  in number.
Post-operative pain scale. | 24 hours postoperative.
  by Visual analogue scale (VAS): (where 0 means no pain- while 100 mm is the worst pain) at 0, 1, 2, 6, 12 and 24 hours.
Intra-operative fentanyl consumption. | Intraoperative (2 hours).
  in micro grams.
Heart rate (HR). | Intraoperative (2 hours), postoperative for 24 hours.
  in beat/minutes, recorded basal, intraoperative: after the block 15 min and 30 min then every 30 minutes till the end of surgery, then postoperative at 0, 1, 2, 6, 12 and 24 hours.
Mean arterial blood pressure (MAP). | Intraoperative (2 hours), postoperative for 24 hours.
  Non invasive mean arterial pressure, in mmHg, recorded intraoperative: basal, after the block at 15 min and 30 min then every 30 minutes till the end of surgery, then postoperative at 0, 1, 2, 6, 12 and 24 hours.
Intra-operative atracurium consumption | Intraoperative (2 hours).
  in milligrams.
The concentration of isoflurane. | Intraoperative (2 hours).
  in percent, recorded after the block every 30 minutes till the end of surgery.
Sensory block assessment. | 1 hour post-operative.
  Define the number of blocked dermatomes at post anesthesia care unit by skin pinprick. sensation at dermatomal distribution.
The block procedural duration. | 30 minutes.
  In minutes.
Post-operative complication rate (nausea, vomiting and headache) | 24 hours postoperative.
  In number.
Assessment of diaphragmatic dysfunction. | 1 hour postoperative.
  Using ultrasound assessment,

CONTACTS AND LOCATIONS:
Overall Officials: Alaa M Mazy, Study Director — Oncology Center, Mansoura University, Egypt.
Locations (1):
- Oncology Center, Mansoura University (OCMU), Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
after publication.
Supporting Information: CSR
Time Frame: 2 years.